CLINICAL TRIAL: NCT00846677
Title: A Randomized, Open-label, Cross-over Study Comparing Two Vitamin D Supplements for Infants: Liquid Versus D-Strips.
Brief Title: Study Comparing Two Vitamin D Supplements for Infants: Liquid Versus D-Strips
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Hope Weiler, Associate Professor, McGill University
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: PLB-D301
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-03

CONDITIONS: Healthy
Keywords: Healthy; Infants; Vitamin D
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Vitamin D quick dissolve strip
  Interventions: Dietary Supplement: Vitamin D, cholecalciferol
- 2 (Active Comparator): Vitamin D syrup
  Interventions: Dietary Supplement: Vitamin D, cholecalciferol

INTERVENTIONS:
Dietary Supplement: Vitamin D, cholecalciferol — Oral Quick Dissolve Strip, 400 IU once per day for 21 days
  Other Names: BabyVita Vitamin D
  Arms: 1
Dietary Supplement: Vitamin D, cholecalciferol — Oral Syrup, 400IU per day for 21 days
  Arms: 2

SUMMARY:
Vitamin D supplementation (400 IU/d) is recommended for all breastfed infants in Canada. Such recommendation is grounded in the fact that the prevalence of rickets in Canada is higher than desirable, likely due to low maternal-fetal transfer and low intakes postpartum.

There is little data about adherence to supplementation in Canada, but one study shows that in primiparous mothers (n=1937) in Quebec, 58.1 % of those exclusively breast-feeding gave their infant vitamin D supplements in the first six months and 62.1 % of those feeding formula did not. For the Canadian situation, it is not clear if the modality of the supplementation is a barrier to providing the supplement. Thus the overall aim of this study is to test a new delivery system for parental preference and infant acceptance compared to a standard vitamin D supplement.

DETAILED DESCRIPTION:
OBJECTIVES

1. To determine parental preference for a new vitamin D delivery system over the standard of care supplement in syrup form.
2. To determine infant acceptance for a new vitamin D delivery system over the standard of care supplement in syrup form.
3. To establish possible barriers to either supplement delivery system being given during infancy.

METHODOLOGY Design: randomized cross-over design, open label. Visit 1 (D1): written consent, demographic survey at first visit, randomize to order of supplement trial to begin with D Strip or syrup drops. obtain infant weight, complete health survey, instruct how to use supplement Call 1 (D4-D6): telephone call to address any questions or concerns, remind of next visit.

Visit 2 (on or around D21): complete survey instrument for first supplement, obtain infant weight, complete health survey, instruct how to use second supplement Call 2: (D25-27): telephone call to address any questions or concerns, remind of next visit.

Visit 3 (on or around D42): complete survey instruments, obtain infant weight; education regarding continued use of vitamin D.

Demographics: Information related to demographics will be obtained at the baseline research visit. This survey (see appendix) includes questions related to parent education, income, and knowledge of vitamin D and prior supplementation practices. This information is important to help understand if parents of all backgrounds accept the supplement delivery systems.

Delivery Systems: Both delivery systems will provide 400 IU of vitamin D3 in accordance with Health Canada's recommendation for all breastfed infants to receive a daily supplement until such dosage can be achieved through other foods (1). The standard delivery system is syrup administered in 1 ml volumes using a dropper. The syrup is typically given in the pockets between the gums and cheeks or slowly on the tongue. The new system is a D Strip that is a small rectangular strip administered on the oral palate (roof of the mouth), inner cheek, or surface of the tongue where it readily adheres and dissolves. Both can be given before or after feeding. The standard liquid supplement will be commercially-available product.

Protocol and Testing: Parents of newborn infants will be asked to participate in the study. In total 50 infants will be studied at baseline beginning at 2 to 4 weeks of age and followed for a total of 6 weeks. At baseline Day 1 (Visit 1) and the beginning of the second study phase a general health assessment questionnaire will be administered. This includes maternal weight and height plus infant weight and overall health of the infant (i.e. any existing illnesses). Should the infant be unwell due to infections such as a common cold at that time, the parent will be asked to begin the study 1 week later provided that the illness has resolved. At Visit 1, parents will be asked demographic information and randomized to either the syrup group or the D Strip group. A registered nurse will show parents how to take the supplement. Then the infant will be weighed if not already done and enough supplement provided for 3 weeks. The first dose of the supplement will then be administered to the infant by the parent in the presence of the nurse. Parents will be informed that a care-call (Call 1) will be made at Day 4 to 6 into the study to establish if they have any questions or concerns. After 3 weeks (i.e. on or around Day 21, but not before the infant has completed 21 days of supplement) the parents and infant will return (Visit 2) to the research site to complete surveys, have the infant weighed and be shown how to administer the other supplement. Again enough supplement will be given and parents informed of a care-call (Call 2) at 4 to 6 days into the supplement trial (i.e. on Day 25-27). The first dose of the supplement will then be administered to the infant by the parent in the presence of the nurse. After 3 weeks (i.e. on or around Day 42, but not before the infant has completed 21 days of supplement) they return for a final visit (Visit 3) to complete surveys (self-administered or with assistance) and have the infant weighed. At this visit, which is the end of study, parents will be given education about the importance of giving their infant vitamin D supplementation until 400 IU can be obtained from food.

Two testing approaches will be used (see appendix) at the end of each study phase. First a validated questionnaire will be used, the medication acceptance scale (MAS), will be used to learn of infant acceptance. The effectiveness and infant acceptance of medications delivered through various modalities has been tested using a MAS designed and validated for pediatric oral liquids (21). This scale uses a point scale generated by observed behavior as related to 4 main areas and has been slightly modified for our use. The second approach will be to administer a parent preference questionnaire using a Likert item response on a scale from 1 to 10.

Compliance Record: To establish compliance with giving daily supplementation three approaches will be taken.

1. Each supplement will be provided in a box with a label fixed to the front upon which parents will initial every dosage given;
2. Parents will be asked for frequency of dosage over each study phase; and
3. Parents will be asked to return remaining supplement at the end of each study phase. Either a count for the D Strip or a weight for the syrup will confirm appropriate number of dosages given.

Compliance will primarily be determined by the returned supplement count. If supplement is not returned, parent recollection of frequency of dosage will be used.

ELIGIBILITY:
Inclusion Criteria:

* Healthy singleton newborn infants born at term age of any racial background.
* Infants may be breastfed or formula fed during the study as is safe since the supplement is 400 IU/d and intakes from breast milk or formula will not exceed 400 IU/d for a theoretical total intake of 800 IU/d that is recommended by the Canadian Pediatric Society.

Exclusion Criteria:

* Infants born prematurely, twins or other multiples.
* Unable to nurse or accept the supplement.
* Congenital malformations.
* Parents not fluent enough in English or French to provide written informed consent.

Ages: 2 Weeks to 4 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2009-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Parental and infant preference for a new vitamin D delivery system over the standard of care supplement in syrup form. | 21 days

SECONDARY OUTCOMES:
Barriers to either supplement delivery system being given during infancy. | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Hope A Weiler, PhD, Principal Investigator — McGill University
Locations (1):
- Mary Emily Clinical Nutrition Research Unit, Sainte-Anne-de-Bellevue, Quebec, Canada

REFERENCES:
- [Derived] Huey SL, Acharya N, Silver A, Sheni R, Yu EA, Pena-Rosas JP, Mehta S. Effects of oral vitamin D supplementation on linear growth and other health outcomes among children under five years of age. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD012875. doi: 10.1002/14651858.CD012875.pub2. PMID 33305842